CLINICAL TRIAL: NCT01740063
Title: Randomized, Double-blind, Placebo-controlled Phase 2B Study on Safety and Therapeutic Efficacy of DAS181 in Adult Subjects With Naturally Acquired Influenza.
Brief Title: Phase 2B Study on Safety and Therapeutic Efficacy of DAS181 in Adult Subjects With Naturally Acquired Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ansun Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAS181-2-04
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DAS181-F02 formulation (Experimental): DAS181 10 mg dose for three days of the F02 formulation
  Interventions: Drug: DAS181-F02 formulation
- DAS181-F04 formulation (Experimental): DAS181 20 mg dose group for three days of the F04 formulation,
  Interventions: Drug: DAS181-F04 formulation
- Placebo (Placebo Comparator): placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DAS181-F02 formulation
  Arms: DAS181-F02 formulation
Drug: DAS181-F04 formulation
  Arms: DAS181-F04 formulation
Drug: Placebo
  Arms: Placebo

SUMMARY:
This protocol will seek to enroll 372 adult otherwise healthy subjects presenting with influenza-like illness (ILI). Subjects will enter the study based on listed inclusion/exclusion criteria, including a positive Rapid Antigen Test (RAT) for influenza virus (IFV).

Subjects will be randomized into one of three treatment groups: a DAS181 30 mg total dose group (DAS181-F02 formulation), a DAS181 60 mg total dose group (DAS181-F04 formulation) or a placebo group.

The modified intent to treat (mITT) analysis set will include subjects with confirmed influenza as documented by qPCR or TCID50. The full analysis set will be used for activity analysis and will include all randomized subjects with baseline and treatment data. Per protocol, the safety analysis sets are described below in statistical methods.

A subpopulation of 60 participants will also have additional PK and Immunogenicity blood samples collected. For this subgroup, PK and Immunogenicity samples will be collected at all study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects in generally good health in the opinion of the investigator as determined by vital signs, medical history, and a physical exam based on medical history.
2. Subjects must be able to verbalize understanding of the consent form, provide written informed consent and verbalize willingness to complete study procedures.
3. Be 18 to 70 years of age (inclusive).
4. Subjects must weigh at least 50 kg and must have a Body Mass Index (BMI) of no greater than 40.00.
5. Febrile, oral temperature ≥100.4°F (≥38.0°C) in combination with symptoms
6. At least one respiratory symptom:

   * Cough
   * Sore throat
   * Wheezing
   * Sneezing
   * Shortness of breath
   * Nasal congestion
   * Earache
   * Pleuritic chest pain
7. At least one constitutional symptom:

   * Headache
   * Myalgia (body aches and pains)
   * Fever or feverish (sweat/chills)
   * Prostration (fatigue, tired, lacking energy)
8. Positive rapid antigen test (RAT) for influenza performed using FDA-cleared and CLIA-waived commercially available rapid antigen test supplied by the sponsor.
9. Blood pressure within normal limits (systolic 90-150 mmHg; diastolic 50-95 mmHg) and heart rate between 45 and 140 beats per minute.
10. Onset of symptoms no more than 48 hours prior to diagnosis.

Note: Time of onset of illness is defined as either:

1. the time when the temperature was first measured as elevated (38 C) OR
2. the time when the subject experienced the presence of at least one symptom, whichever occurs first 11. Female subjects must be post-menopausal (one year or greater without menses), surgically incapable of childbearing, or practicing two effective methods of birth control. Acceptable methods may include intrauterine device, spermicide, barrier and hormonal contraception. A female subject must agree to practice an acceptable method of birth control during the study period. All female subjects regardless of menopausal status or surgical history must have had a negative urine pregnancy test during the screening visit and prior to dosing.

12. Male subjects must agree to use medically accepted form of contraception during the study period.

Exclusion Criteria:

1. Have received any investigational drug or investigational vaccine within 8 weeks prior to study drug dosing.
2. Have had a serious adverse reaction or previous episode of anaphylaxis related to any drug.
3. Have received blood products within 6 months of study enrollment.
4. Have concurrent cystic fibrosis or emphysema.
5. Have sickle cell disease.
6. Known IGE mediated allergic response to lactose (not lactose intolerance).
7. Any history of congenital or acquired bleeding abnormalities.
8. Existence of any surgical, medical, or laboratory condition that, in the judgment of the clinical investigator, might interfere with the safety, distribution, metabolism or excretion of the drug.
9. Use of antiviral influenza medications within 10 days prior to screening (Subjects will be prohibited from taking antiviral influenza medications during the course of the trial).
10. Current clinical evidence of a recognized or suspected uncontrolled non-influenza infectious illness with onset prior to screening.
11. Known hypersensitivity to DAS181.
12. Women who are pregnant (urine pregnancy test), who are attempting to become pregnant, or who are breast-feeding.
13. Uncontrolled seizure disorder or history of seizure activity within 12 months prior to study participation.
14. Any significant findings in the subject's medical history or physical examination that, in the opinion of the investigator, would affect subject safety or compliance with the dosing schedule.
15. Subjects with history of asthma or chronic obstructive pulmonary disease (COPD) requiring the use of acute or chronic medication in the past 3 years.
16. Subjects with acute diagnosis of a chronic medical condition within the last 3 months.
17. Subjects with a chronic medical condition that have initiated or changed dosing or regimen of prescription medications to treat the chronic medical condition within the last 3 months. (Any changes in chronic medications during the 28 day enrollment period will be captured in the source documentation under concomitant medications).
18. Subjects with current or previous history of the following: systemic disorders, immunological disorders, hepatitis B virus (HBV), hepatitis C virus (HCV) or cirrhosis, transplant recipients, or other immunosuppressive illness.
19. Subjects with cancer or history of hematologic malignancy. Cancer is defined as any active neoplastic diseases excluding noninvasive basal cell carcinoma.
20. Subjects who have had or are scheduled to have surgery within 30 days of initiation of the study.
21. Subjects who have donated or lost more than 500 mL of blood in the two months prior to screening.
22. Psychiatric or cognitive illness or recreational drug/alcohol use that, in the opinion of the principal investigator, would affect subject safety and/or compliance.
23. Family members of site staff directly involved in study conduct are excluded from study participation.
24. Subjects with an oxygen saturation (Sa02) level of <92% as measured by pulse oximeter.
25. Subjects with a modified CURB-65 score of 2 or higher.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2012-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with Unacceptable Serious Adverse Events due to safety and toxicity Safety and toxicity profile: Unacceptable Serious Adverse Events Safety and toxicity profile: Unacceptable Serious Adverse Events | Participants will be followed (up to one year) for the duration of the study and outcome measure will be reviewed at the end of study. The expected end of study is Sept. 2013.
  Because of the possibility of unacceptable or excessive defined serious adverse events during the treatment period or the study enrollment period, a stopping rule for safety/tolerability has been introduced in the design.
  The following two stopping rule criteria will initiate an ad hoc DSMB data evaluation.
  * 5% with a related SAE post-dose Day 1 through Day 28 , or
  * 15% with related DAIDS toxicity Grade 3 and 4 laboratory abnormalities post-dose Day 1 through Day 28
    * Grade 3 laboratory abnormalities in hematology or serum chemistry, excluding absolute neutrophils and absolute lymphocytes.
    * Grade 4 laboratory abnormalities in hematology or serum chemistry including absolute neutrophils and absolute lymphocytes
  Changes (absolute and percent) from baseline in influenza viral load from Day 1 to Day 2 as measured by quantitative polymerase chain reaction (qPCR) from pharyngeal wash and nasal wash samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Nexbio, San Diego, California, United States